CLINICAL TRIAL: NCT00437086
Title: A Prospective Open-Label Pilot Trial of PS-341 (Bortezomib; VELCADE) for the Therapy of Symptomatic Advanced Myeloproliferative Disorders
Brief Title: Bortezomib in Treating Patients With Advanced Myeloproliferative Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000529906; P30CA015083 (NIH); MC0486 (Other: Mayo Clinic Cancer Center); 695-05 (Other: Mayo Clinic IRB); VEL-04-107 (Other: MPI)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia
Keywords: chronic myelomonocytic leukemia; primary myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Leukemia, Myelomonocytic, Chronic; Primary Myelofibrosis | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PS-341 (Experimental): Designed to assess the toxicity and pilot response of PS-341 in patients with advanced myeloproliferative diseases.
  Interventions: Drug: PS-341

INTERVENTIONS:
Drug: PS-341 — 1.6 mg/m2 by IV; 4 out of 5 weeks
  Other Names: Bortezomib, Velcade, MLN-341, LDP-341

SUMMARY:
RATIONALE: Bortezomib may stop the growth of abnormal cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the abnormal cells.

PURPOSE: This clinical trial is studying the side effects and how well bortezomib works in treating patients with advanced myeloproliferative disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of bortezomib in patients with symptomatic advanced myeloproliferative disorders (i.e., myelofibrosis with myeloid metaplasia, chronic myelomonocytic leukemia, or FIP1LI-PDGFRA-negative mast cell disease).
* Determine the safety of this drug when administered on a modified schedule in these patients.

Secondary

* Determine the effect of this drug on bone marrow cellularity, tryptase-positive mast cells, reticulin fibrosis, osteosclerosis, and angiogenesis in responding patients

OUTLINE: This is a prospective, open-label, pilot, multicenter study. Patients are stratified according to disease (systemic mast cell disease vs chronic myelomonocytic leukemia vs myelofibrosis with myeloid metaplasia).

Patients receive bortezomib IV weekly for 4 weeks. Treatment repeats every 5 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a response (complete remission, partial remission, or minimal remission) after 2 courses may receive an additional 6 courses of therapy. Patients who achieve stable disease with acceptable toxicities after 2 courses receive bortezomib IV at a higher dose twice weekly for 2 weeks. Treatment with a higher dose of bortezomib repeats every 3 weeks for up to 6 courses.

Patients who are responders undergo bone marrow aspirate or biopsy and peripheral blood collection for evaluation of bone marrow cellularity, tryptase-positive mast cells, reticulin fibrosis, osteosclerosis, and angiogenesis by fluorescent in situ hybridization (FISH), immunohistochemistry, and other immunological laboratory methods.

After completion of study therapy, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced myeloproliferative disorder, including 1 of the following subtypes:

  * Myelofibrosis with myeloid metaplasia defined by the following criteria:

    * Evaluable or symptomatic disease as evidenced by ≥ 1 of the following:

      * Anemia, defined as hemoglobin < 10 g/dL OR erythrocyte-transfusion dependence, defined as requiring 1 transfusion within the past 8 weeks
      * Symptomatic palpable splenomegaly (palpable hepatomegaly is acceptable if previously splenectomized) requiring treatment* NOTE: *Subjective but painful enough to mandate intervention
  * Chronic myelomonocytic leukemia (CMML) defined by the following criteria:

    * Absence of an imatinib mesylate-sensitive molecular abnormality for CMML (i.e., t[5;12], t[5;10], t[1;5], and t[5;7]) confirmed by fluorescent in situ hybridization (FISH) or standard cytogenetic bone marrow analysis within the past 18 months
    * Symptomatic disease as evidenced by ≥ 1 of the following:

      * Anemia, defined as hemoglobin < 10 g/dL OR erythrocyte-transfusion dependence, defined as requiring 1 transfusion within the past 8 weeks
      * Palpable splenomegaly (palpable hepatomegaly is acceptable if previously splenectomized) requiring treatment* NOTE: *Subjective but painful enough to mandate intervention
      * Leukocytosis associated with ascites, serositis, pleural effusions, vasculitis, or other overt manifestation
  * Systemic mast cell disease defined by the following criteria:

    * Absence of the FIP1LI-PDGFRA mutation as confirmed by FISH
    * Evaluable and symptomatic disease requiring therapy, as evidenced by involvement with organs other than skin (i.e., heart, bowel, peripheral blood, liver/spleen, or marrow)
    * Debilitating mast cell mediator symptoms not responsive to standard therapy such as antihistamines
* Absence of t(9;22) translocation as confirmed by FISH or standard cytogenetic peripheral blood or marrow analysis at any prior time point

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Not incarcerated in a municipal, county, state, or federal prison
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Total or direct bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 3 times upper limit of normal (unless clinically attributed to hepatic extramedullary hematopoiesis)
* No baseline peripheral or autonomic neuropathy ≥ grade 2
* No other condition or laboratory abnormality that would place the patient at unacceptable risk or confound the ability to interpret study data
* No hypersensitivity to boron, mannitol, or bortezomib
* No myocardial infarction within the past 6 months
* No New York Hospital Association class III-IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmia
* No evidence of acute ischemia or active conduction system abnormality by ECG

  * ECG screening abnormalities must be documented as not medically relevant
* No other serious medical or psychiatric illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

* At least 14 days since prior chemotherapy (e.g., interferon alfa, anagrelide, or other myelosuppressive agent) or any other experimental therapy
* At least 14 days since prior growth factors
* At least 14 days since prior systemic use of corticosteroids
* More than 14 days since prior investigational drugs
* Concurrent hydroxyurea allowed for ≤ 14 days during study therapy if clinically indicated for extreme leukocytosis control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Number and severity of toxicities as assessed by NCI CTCAE v3.0 | 40 weeks
Proportion of patients who show treatment success, as defined by anemia, spleen, bone marrow, or constitutional symptoms' response (complete, partial, major, or minor response) | 40 weeks

SECONDARY OUTCOMES:
Effects of treatment, in terms of changes in bone marrow cellularity, tryptase-positive mast cells, reticulin fibrosis, osteosclerosis, and angiogenesis, in responding patients | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ruben A. Mesa, M.D., Study Chair — Mayo Clinic; Candido E. Rivera, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas